CLINICAL TRIAL: NCT02444962
Title: Safe and Easy Application of BioComp Implants for Prosthetic Reconstruction of Craniofacial Defects
Brief Title: BioComp Implants in Anaplastology - Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC142065
Record Dates: First submitted 2014-12-22; First posted 2015-05-15 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Prostheses and Implants; Craniofacial Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAVD implant (Experimental)
  Interventions: Device: HAVD-implant

INTERVENTIONS:
Device: HAVD-implant — hydroxy-apatite coated, acid etched implant for extra oral use to reconstruct craniofacial defects with an episthesis

SUMMARY:
At the department of Cranio-Maxillofacial Surgery, Maastricht University Medical Center (MUMC) the routine procedure after ablation of the nose, ear or eye is reconstruction with an episthesis. Retention can be achieved using adhesives, undercuts or bone implants. Implant based episthesis are now commonly used because of the good retention and episthesis stability. This results in a better patient quality of life.

Today we use machined surface implants in the craniofacial region of different brands. Each system has its own instruments and application method. To enhance the clinical usability, we are searching for one system for all extra-oral implant regions.

Furthermore, implant patients may be compromised by aging, diseases, smoking, medication and radiation therapy, which can affect the bone healing process. In these cases, implants are known to have higher failure rates compared to the application in healthy cases. Therefore implants with biomechanical surface modifications, such as the HAVD implants of BioComp, may have a positive effect on osseointegration, resulting in higher success rates in the compromised patient.

The aim of this pilot study is to collect information about the functionality and safety of a surface treated implant system (HAVD, BioComp) for episthetic reconstruction after ablative surgery in the nasal, orbital and auricular region for a potential future RCT.

ELIGIBILITY:
Inclusion Criteria:

* In need of an auricular, nasal or orbital episthesis
* Be able to maintain a good personal hygiene

Exclusion Criteria:

* Contraindications for general anesthesia
* DEmentia or other psychiatric disorders/ unable to maintain a good personal hygiene
* Poor personal hygiene
* Pregnancy
* Acute infection
* Immunosuppression
* Compromised by medication
* Local irradiation >50Gray

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in implant stability as measured by the Osstell implant stability meter at one year | one year

SECONDARY OUTCOMES:
redness/irritation of the skin | baseline
redness/irritation of the skin | 12 weeks after implant placement
redness/irritation of the skin | 26 weeks after implant placement
redness/irritation of the skin | 52 weeks after implant placement
Implant survival | 52 weeks after implant placement
Clinical ease of use | Directly after implant placement (0)
  Opinion of the surgeon about the easiness of use of the implant system, scored by a questionnaire.
Patient satisfaction as measured by a VAS scoring system | 26 weeks after implant placement
  Patient satisfaction scored by a self made questionnaire
Patient satisfaction as measured by a VAS scoring system | 52 weeks after implant placement
  Patient satisfaction scored by a self made questionnaire
Quality of life a measured by a VAS scoring system | 52 weeks after implant placement
  Quality of life scored by a self made questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter AW Kessler, Prof. Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands